CLINICAL TRIAL: NCT00490230
Title: Assessment of Cutaneous Leishmaniasis Scar (Caused by Leishmania Major) for Cosmetic Outcome After Treatment With WR279396 (Paromomycin/Gentamicin Cream in Vehicle) Versus a No Treatment Control Group (Natural Healing)
Brief Title: Cosmetic Outcome of Leishmaniasis Scar After WR279396 Application
Acronym: SCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: WRAIR 1303
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Cutaneous Leishmaniasis; Scar
Keywords: Paromomycin; Gentamicin
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- WR 279,396 (Experimental): CL lesions treated with WR 279396
  Interventions: Drug: WR 279396
- Natural Healing (No Intervention): CL lesions healed naturally
- vehicle control (Placebo Comparator): CL lesions were treated with the vehicle alone
  Interventions: Drug: WR 279396

INTERVENTIONS:
Drug: WR 279396
  Arms: WR 279,396; vehicle control

SUMMARY:
Primary Objectives:

Assess whether CL (caused by Leishmaniasis major) lesions treated with WR279396 improved the cosmetic outcome compared with no treatment (natural healing)

DETAILED DESCRIPTION:
Secondary Objectives

1. Evaluate the cosmetic outcome of CL lesions treated with "vehicle" compared with no treatment (natural healing)
2. Evaluate the cosmetic outcome of CL lesions treated with "vehicle" compared with WR279396

   * To determine whether CL lesions treated with vehicle improves the cosmetic outcome (compared with natural healing)
   * To determine whether CL lesions treated with vehicle alone provides a cosmetic outcome similar to WR279396

ELIGIBILITY:
Inclusion Criteria:

* Included are volunteers who participated in WRAIR 813 (HSRRB Log # 9768.1) and those who participated in another CL study in/around the WRAIR 813 study site who had been assigned to a "no-treatment" (natural healing) arm. All volunteers will have had documented CL in the past that were treated with WR279396, vehicle, or no treatment (natural history), have signed informed consent, and are willing to comply with study assessments; age range: 5 to 75 years old.
* For study subjects who were enrolled in WRAIR 813 in 2004 (WR279396 or vehicle treated):

  * Written informed consent obtained from the subject or guardian
  * Willing to meet the requirements of the single clinic visit
  * Prior data in the clinical site data base documenting a diagnosis of CL
  * Each lesion for inclusion in this study conforms to WRAIR 813: ³ 1 cm in diameter and was primarily ulcerative (i.e., not verrucous or nodular)
  * The index lesion and others to be scored were proven parasitologically by Giemsa slide smear
  * CL scars documented to be > 360 days old (clock starts at time of diagnosis)
  * No treatment of the lesions other than that received in the previous protocol
* Study subjects from the earlier studies to serve as "no treatment" controls:

  * Written informed consent obtained from the subject or guardian
  * Willing to meet the requirements of the single clinic visit
  * Same age range as WRAIR 813: 5-75 years old at time of diagnosis
  * Prior data in the clinical site data base documenting a diagnosis of CL, and that the volunteer was assigned to the "no treatment" group
  * Each lesion for inclusion in this study will conform to WRAIR 813: at the time of diagnosis, ≥1 cm in diameter and described as primarily ulcerative (i.e., not verrucous or nodular)
  * At least 1 lesion that was proven parasitologically by Giemsa slide smear for inclusion in the earlier study.
  * CL scars documented to be > 360 days old (clock starts at time of diagnosis)
  * Never received any treatment of the lesions (natural healing) or applied any medication, such as herbal medication
  * Lesions present on the trunk or extremities, to match the WRAIR 813 study volunteers (no facial lesions were treated in the 2004 study)

Exclusion Criteria:

* Potential volunteers without a prior documented diagnosis of CL

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Cosmetic outcome based on modified Vancouver Scar Score (mVSS) | Day 360 or greater
  The primary cosmetic outcome measure is the Clinical Scar Rating, based on a modified Vancouver Scar Score (mVSS). The primary efficacy endpoint is the percent of persons judged to have either a "superior (no scar)" or "excellent" rating (see below).

CONTACTS AND LOCATIONS:
Overall Officials: COL Doug Walsh, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Institute Pasteur de Tunis, Tunis, Tunisia